CLINICAL TRIAL: NCT05588401
Title: Phase 1/2a First-in-human Trial Evaluating Autologous Gene-edited Muscle Stem Cells in Limb Girdle Muscular Dystrophies (GenPHSats-bASKet)
Brief Title: Evaluating Safety and Efficacy of Autologous Gene-edited Muscle Stem Cells (GenPHSats-bASKet)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Simone Spuler, MD (Other)
Responsible Party: Sponsor-Investigator, Simone Spuler, MD, Clinical Professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: bASKet
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: LGMD
MeSH Terms: interventions — Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GenPHSat safety injection and GenPHSat efficacy injection (Experimental): Initial intervention with six injections into the left biceps. A second intervention with 36 injections into the right biceps.
  Interventions: Biological: GenPHSat injection (Safety); Biological: GenPHSat injection (Efficacy); Other: Muscle Biopsy (Safety)

INTERVENTIONS:
Biological: GenPHSat injection (Safety) — Participants receive gene edited primary human muscle stem cells (GenPHsat) injection in the left biceps muscle.
Biological: GenPHSat injection (Efficacy) — Participants receive gene edited primary human muscle stem cells (GenPHsat) injection in the right biceps muscle.
Other: Muscle Biopsy (Safety) — Participants undergo muscle biopsy 3 month after safety GenPHSat injection.

SUMMARY:
This study is an investigator initiated first-in-human interventional open label phase 1/2a clinical trial investigating an ATMP in the orphan disease LGMD to evaluate safety and efficacy.

DETAILED DESCRIPTION:
This trial is directed towards a first-in-human application of GenPHSats; gene edited primary human satellite cell derived muscle stem cells as a new Advanced Therapy Medicinal Product (ATMP) in a phase 1/2a clinical trial with Gene edited PHSats (GenPHSats) initiating healthy muscle development in patients with LGDM. The trial is set up to verify if GenPHSats can provide an therapy option for LGDM patients as there is currently no therapy available. The GenPHSats are an autologous product comprised of primary human satellite cell derived muscle stem cells obtained from the patient's own muscle tissue and gene edited in vitro prior to transplantation.

ELIGIBILITY:
Inclusion Criteria:

* LGDM diagnosed,
* Identified gene defect location and gene editing proved feasible,
* Age ≥14 years,
* Patient in treatment in the department at Charité, Universitätsmedizin Berlin, Muscle Research Unit and Outpatient Clinic for Muscle Disorders,
* Signed informed consent

Exclusion Criteria:

* Acute or chronic inflammatory local or systemic disease
* Coagulation disorder
* Known complications due to local anesthesia,
* Congenital heart defect, cardiac arrhythmia,
* Pathology of the airways such as micrognathia
* Pierre Robin Sequence
* Central hypoventilation syndrome/Ondine syndrome
* Significant other medical or psychiatric illness
* Positive serology for HIV and/or hepatitis A, B, C
* Pregnant or lactating women
* Known allergic reaction to constituents of the cryopreservation medium

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 1 year
  Characterization of type, incidence, severity, duration, reversibility, treatability of adverse events recorded at least at visit 1, 2, 3 and 4 (end of trial).

SECONDARY OUTCOMES:
Rate of muscle biopsy post-injection structure | 3 month post injection
  The muscle biopsy taken and stained to visualize muscle biopsy structure after 3 month post injection.

OTHER OUTCOMES:
Rate of Muscle force | Until 6 month post injection
  Muscle force measurement data taken at screening (baseline), visit 1, 2, 3 and 4 (end of trial).
Rate of Blood CK | Until 6 month post injection
  CK blood determination at screening (baseline), visit 1, 2, 3 and 4 (end of trial).

CONTACTS AND LOCATIONS:
Overall Officials: Simone Spuler, Prof Dr med, Study Chair — Charite Universitätsmedizin Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided